CLINICAL TRIAL: NCT01976923
Title: Pre-Operative Intravitreal Bevacizumab for Tractional Retinal Detachment Secondary to Proliferative Diabetic Retinopathy: Results of the Pan-American Collaborative Retina Study (PACORES) Group
Brief Title: Pre-Operative Intravitreal Bevacizumab for Tractional Retinal Detachment Secondary to Proliferative Diabetic Retinopathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: J. Fernando Arevalo, MD FACS (Other Government)
Collaborators: Pan American Collaborative Retina Study Group (Network)
Responsible Party: Sponsor-Investigator, J. Fernando Arevalo, MD FACS, Chief of Vitreoretina Division, King Khaled Eye Specialist Hospital
Organization: King Khaled Eye Specialist Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1338-P
Record Dates: First submitted 2013-10-25; First posted 2013-11-06 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Tractional Retinal Detachment Secondary to Proliferative Diabetic Retinopathy
Keywords: Intravitreal Bevacizumab; Tractional Retinal Detachment; Proliferative Diabetic Retinopathy; Small gauge pars plana vitrectomy; Intraoperative bleeding; Post-operative vitreous hemorrhage; Visual acuity
MeSH Terms: conditions — Blood Loss, Surgical

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Study arm (Active Comparator): Intravitreal bevacizumab Small-gauge pars plana vitrectomy
  Interventions: Drug: Intravitreal bevacizumab; Procedure: Small-gauge pars plana vitrectomy
- Control arm (Sham Comparator): Small-gauge pars plana vitrectomy
  Interventions: Procedure: Small-gauge pars plana vitrectomy

INTERVENTIONS:
Drug: Intravitreal bevacizumab — A sterile lid speculum is used to separate the lids. A subconjunctival injection of 1% lidocaine is applied to the inferotemporal quadrant. A 5% povidone iodine solution is used to disinfect the entire conjunctival surface. 1.25 mg / 0.05 mL of bevacizumab is injected using a 30-gauge needle inserted through the inferotemporal pars plana 3.5 mm from the limbus.
  Arms: Study arm
Procedure: Small-gauge pars plana vitrectomy

SUMMARY:
The purpose of this is study is to assess the efficacy of pre-operative intravitreal bevacizumab (IVB) (Genentech, South San Francisco CA) in improving visual acuity, reducing operative time, complications, intra-operative and post-operative hemorrhage following small gauge pars plana vitrectomy (PPV) (23-gauge, 25-gauge or 27-gauge ) compared to small gauge PPV (23-gauge, 25-gauge or 27-gauge) alone in eyes with tractional retinal detachment (TRD) secondary to proliferative diabetic retinopathy (PDR). Hypothesis: Preoperative IVB may be beneficial for membrane dissection in diabetic tractional retinal detachment with minimally invasive vitreoretinal surgery (23-gauge transconjunctival sutureless vitrectomy [TSV]). In addition, post-operative rebleeding may be decreased.

DETAILED DESCRIPTION:
This will be a prospective, randomized, active-controlled study of 224 eyes of patients with the diagnosis of TRD secondary to PDR. Participants will be screened for eligibility. Eligible patients will be examined at baseline to determine their ocular condition and randomized into 2 arms. Patients will be randomized in a 1:1 ratio to the study arm.

1. Control arm: PPV without pre-operative bevacizumab (Sham injection).
2. Study arm: Pre-operative bevacizumab (3-5 days) before PPV.

In the study arm, an intravitreal bevacizumab injection at a dose of 1.25 µg/0.05 mL will be scheduled 3 to 5 days before minimally invasive vitreoretinal surgery (MIVS).

The purpose of the current study is to determine the effectiveness and safety of an intravitreal injection of 1.25 mg of bevacizumab as a pre-operative adjunct to PPV in eyes with TRD secondary to PDR.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years with proliferative diabetic retinopathy (PDR) and tractional retinal detachment (TRD) threatening or involving the fovea.
2. Diagnosis of diabetes mellitus (type 1 or type 2)
3. At least one eye meets the study eye criteria
4. One eye per patient will be included
5. Able and willing to provide informed consent prior to any study-related procedures
6. Best corrected visual acuity 20/40 or less
7. Willing and able to comply with clinic visits and study-related procedures
8. U.S. patients will be required to have a Health Insurance Portability and Accountability Act (HIPAA) authorization; in other countries, as applicable according to national laws

Exclusion Criteria:

Ocular Exclusion Criteria

The following exclusions apply to the study eye only (i.e., they may be present for the non-study eye):

1. TRD is considered to be due to a cause other than diabetes.
2. An ocular condition is present such that, in the opinion of the investigator, visual acuity loss would not improve from resolution of TRD (e.g., foveal atrophy, pigment abnormalities, dense subfoveal hard exudates, nonretinal condition, optic atrophy).
3. An ocular condition is present (other than diabetes) that, in the opinion of the investigator, might affect retinal status or alter visual acuity during the course of the study (e.g., retinal vein occlusion, uveitis or other ocular inflammatory disease, glaucoma, etc.)
4. History of treatment for diabetic macular edema or diabetic retinopathy at any time in the past 4 months with anti-vascular endothelial growth factor (VEGF) drugs.
5. History of major ocular surgery (including vitrectomy, cataract extraction, scleral buckle, any intraocular surgery, etc.) within prior 4 months of randomization.
6. History of neodymium-doped yttrium aluminium garnet (YAG) capsulotomy performed within 2 months prior to randomization.
7. Intraocular pressure >= 25 mmHg.
8. Exam evidence of external ocular infection, including conjunctivitis, chalazion, or significant blepharitis
9. An ocular condition is present (other than diabetes) that, in the opinion of the investigator, might affect retinal status or including hypertension, cardiovascular disease, and glycemic control.

Systemic Exclusion Criteria

A participant is not eligible if any of the following exclusion criteria are present:

1. Significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant.
2. A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including hypertension, cardiovascular disease, and glycemic control).
3. Participation in an investigational trial within 30 days of randomization that involved treatment with any drug that has not received regulatory approval at the time of study entry.
4. Known allergy to any component of the study drug.
5. Blood pressure > 180/110 mmHg (systolic above 180 or diastolic above 110).
6. Major surgery within 28 days prior to randomization or major surgery planned during the next 6 months.
7. Myocardial infarction, other cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 4 months prior to randomization.
8. Systemic anti-VEGF or VEGF treatment within 4 months prior to randomization.
9. For women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next 12 months.
10. Participant is expecting to move out of the area of the clinical center to an area not covered by another clinical center during the first 12 months of the study.
11. Participation in an investigational trial within 30 days of randomization that involved treatment with any drug that has not received regulatory approval at the time of study entry.
12. Known allergy to any component of the study drug.
13. Blood pressure > 180/110 mmHg (systolic above 180 or diastolic above 110).
14. Major surgery within 28 days prior to randomization or major surgery planned during the next 6 months.
15. Myocardial infarction, other cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 4 months prior to randomization.
16. Systemic anti-VEGF or VEGF treatment within 4 months prior to randomization.
17. For women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next 12 months.
18. Participant is expecting to move out of the area of the clinical center to an area not covered by another clinical center during the first 12 months of the study.
19. History of blood diseases associated with abnormal coagulation.
20. Anti-coagulant therapy (warfarin or heparin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2013-11; Primary Completion 2018-07 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Intraoperative bleeding | 12 months
Total surgical time | 12 months
Post-operative vitreous hemorrhage | 12 months
  Early (<1 month) and late (≥ 1 month) post-operative vitreous hemorrhage (VH) (Yes or No)
Visual acuity change | 12 months
  Mean change in best-corrected visual acuity (BCVA) at 12 months

SECONDARY OUTCOMES:
Number of endodiathermy applications | 12 months
Intraoperative breaks | 12 months
Change in central macular thickness | 12 months
Proportion of eyes gaining at least 15 letters of BCVA | 12 months

OTHER OUTCOMES:
Molecules in the vitreous humor and epiretinal membranes | 12 months
  We would now like to examine molecules in the vitreous humor and epiretinal membranes to gain insight and better assess the efficacy and outcomes of pre-operative intravitreal bevacizumab.

CONTACTS AND LOCATIONS:
Locations (1):
- King Khaled Eye Specialist Hospital, Riyadh, Saudi Arabia

REFERENCES:
- [Background] Arevalo JF, Sanchez JG, Saldarriaga L, Berrocal MH, Fromow-Guerra J, Morales-Canton V, Wu L, Maia M, Saravia MJ, Bareno J; Pan American Collaborative Retina Study Group. Retinal detachment after bevacizumab. Ophthalmology. 2011 Nov;118(11):2304.e3-7. doi: 10.1016/j.ophtha.2011.05.015. No abstract available. PMID 22047908
- [Background] Arevalo JF, Sanchez JG, Lasave AF, Wu L, Maia M, Bonafonte S, Brito M, Alezzandrini AA, Restrepo N, Berrocal MH, Saravia M, Farah ME, Fromow-Guerra J, Morales-Canton V. Intravitreal Bevacizumab (Avastin) for Diabetic Retinopathy: The 2010 GLADAOF Lecture. J Ophthalmol. 2011;2011:584238. doi: 10.1155/2011/584238. Epub 2011 Mar 30. PMID 21584260
- [Background] Arevalo JF, Garcia-Amaris RA. Intravitreal bevacizumab for diabetic retinopathy. Curr Diabetes Rev. 2009 Feb;5(1):39-46. doi: 10.2174/157339909787314121. PMID 19199897
- [Background] Arevalo JF, Maia M, Flynn HW Jr, Saravia M, Avery RL, Wu L, Eid Farah M, Pieramici DJ, Berrocal MH, Sanchez JG. Tractional retinal detachment following intravitreal bevacizumab (Avastin) in patients with severe proliferative diabetic retinopathy. Br J Ophthalmol. 2008 Feb;92(2):213-6. doi: 10.1136/bjo.2007.127142. Epub 2007 Oct 26. PMID 17965108